CLINICAL TRIAL: NCT00563797
Title: Mecamylamine for the Treatment of Patients With Depression and Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0705002629
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Alcohol Dependence; Depression
Keywords: treatment; alcohol dependence; depression; mecamylamine
MeSH Terms: conditions — Alcoholism; Depression | interventions — Mecamylamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mecamylamine (Experimental): Mecamylamine is a noncompetitive, high-affinity nAChR antagonist with low selectivity for the alpha-7 receptor. Those receiving mecamylamine started at 2.5mg once daily (second dose was placebo). The dose was increased to 5.0 mg twice daily over 3 weeks.
  Interventions: Drug: Mecamylamine
- Placebo (Placebo Comparator): Placebo capsules were prepared by the pharmacy and were identical in size and color to the medication capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mecamylamine — mecamylamine 10mg/day for 12 weeks
  Arms: Mecamylamine
Drug: Placebo — Placebo pill
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy of mecamylamine (MEC, 10 mg/day) versus placebo in reducing depressive and alcohol symptoms in patients with depression and co-morbid alcohol dependence. The researchers hypothesize that MEC will significantly reduce depressive symptoms and decrease alcohol consumption compared to placebo in patients with depression and alcohol dependence who are on a stable dose of a selective serotonin reuptake inhibitor (SSRI).

DETAILED DESCRIPTION:
Depression with co-morbid alcohol dependence is very prevalent and it is very costly to treat. The co occurrence of the two disorders leads to greater severity and worse long-term outcome, including suicide. Although a number of treatment strategies have been implemented for depressed patients with alcohol dependence the controversy concerning best treatment options for those patients persists.

The clinical relationship between depression and alcohol dependence suggests some common mechanism underlying both disorders. It has been hypothesized that medications that block presynaptic nAChR may be effective in the treatment of alcoholism and depression. Mecamylamine (Inversine ®) is a noncompetitive, high affinity nAChR antagonist with low selectivity for the alpha-7 receptor. Mecamylamine has never been investigated as an effective adjunct treatment for dually diagnosed patients with depression and alcohol dependence. Methods: Thirty participants with a current diagnosis of depression and alcohol dependence will be recruited for this 12-week treatment study. Fifteen participants will be randomized to mecamylamine and fifteen to placebo. Participants will be included in the study if: they meet current DSM-IV criteria for Major Depression and Alcohol Dependence and have been on a stable SSRI dose for 2 weeks. All participants will come weekly to take their medications and complete weekly assessments. Weekly assessments will consist of questioners that will assess depressive symptoms and alcohol consumption over the entire treatment period. Significance: This study is the first to evaluate the efficacy of mecamylamine as an augmenting agent for treatment of depression and alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with the DSM-IV diagnosis of Major Depression (MD) and Alcohol Dependence (AD) (using the SCID).
2. Individuals who have been on a stable SSRI dose for 2 weeks.
3. Smokers and non-smokers (smokers are defined as smoking more than 5 cigarettes per day).
4. Individuals who have a history of substance dependence (other than alcohol, tobacco and cocaine) but have not met criteria for substance dependence in the past 30 days will be included (using the SCID).
5. Women of childbearing potential must have a negative pregnancy test and use an acceptable method of contraception.
6. Individuals who are able to participate psychologically and physically; give informed consent; complete the assessments; take the study medication; and otherwise participate in the trial. A post-consent test will be given to assess patient's capacity to give informed consent.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Patients may not be taking medications thought to influence drinking behavior, including: acamprosate, disulfiram, naltrexone, or ondansetron.
3. Patients with significant underlying medical conditions, such as cerebral, renal, thyroid, hepatic or cardiac pathology, which in the opinion of the physician would preclude the patient from fully cooperating or be of potential harm during the course of the study.
4. Patients with a history of glaucoma, prostatic hypertrophy, urethral obstruction, cerebral arteriosclerosis, pyloric stenosis, or a history of hypersensitivity to mecamylamine.
5. Patients who meet current SCID criteria for the following major Axis I diagnosis (Posttraumatic Stress Disorders (PTSD), Bipolar Disorders, Schizophrenia and Schizophrenia-type Disorders).
6. Patients with a current unstable medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology (LFT more than 5 times normal, abnormal BUN and creatinine, and unmanaged hypertension with BP higher than 200/120).
7. Patients on pharmacological treatments for alcohol and/or nicotine dependence. (8) Patients taking bethanechol. (9) Patients at risk for suicide.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ralevski, Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 284 subjects were assessed for eligibility, but 263 were excluded because they did not meet inclusion criteria or did not want to participate.
Period: Overall Study
Arm/Group | Mecamylamine | Placebo
Started | 11 | 10
Received Allocated Intervention | 11 | 10
Follow-Up | 11 | 10
Completed | 4 | 8
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 7 | 2

BASELINE CHARACTERISTICS:
Population: Participants were included in the study if they met criteria for major depression and alcohol dependence, had been on a stable antidepressant dose for 2 weeks, and were either smokers or nonsmokers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mecamylamine | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.91 (8.43) | 48.20 (9.84) | 49.62 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 7 | 9 | 16
  African American | 4 | 1 | 5
Drinks per drinking day [Mean (Standard Deviation); unit: drinks per day] | 13.56 (8.27) | 9.32 (8.99) | 11.54 (8.68)
Drinking days, past 30 [Mean (Standard Deviation); unit: drinking days] | 22.55 (7.50) | 22.10 (8.57) | 22.33 (7.83)
Heavy drinking days, past 30 [Mean (Standard Deviation); unit: days] — Heavy drinking days is defined as 5 drinks on a single occasion for men and 4 for women
  days | 21.73 (7.38) | 18.00 (11.62) | 19.95 (9.57)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes] | 13.6 (7.8) | 16.6 (4.50) | 14.9 (6.60)
Total Alcohol Dependence Scale (ADS) score [Mean (Standard Deviation); unit: units on a scale] — The Alcohol Dependence Scale is made of 25 items that cover alcohol withdrawal symptoms, impaired control over drinking, awareness of a compulsion to drink, increased tolerance to alcohol, and salience of drink-seeking behavior. The scale can range from 0 to 47. The higher the value the greater the dependence. A score of 9 or more is highly predictive of DSM diagnosis of alcohol dependence. More specifically, a score from 1-13 indicates low dependence, 14-21 indicates intermediate, 22-30 indicates substantial, and 31-47 severe level of alcohol dependence.
  units on a scale | 17.70 (10.34) | 21.7 (9.72) | 19.70 (9.98)
Depression HAMD [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale (HAM-D) has proven useful for many years as a way of determining a patient's level of depression before, during, and after treatment. It should be administered by a clinician experienced in working with psychiatric patients.
  Although the HAM-D form lists 21 items, the scoring is based on the first 17. It generally takes 15-20 minutes to complete the interview and score the results. The Scale ranges from 0 (normal) to >23 (Very Severe Depression)
  units on a scale | 13.64 (5.43) | 12.90 (2.93) | 13.29 (4.32)
Smoking Status [Number; unit: participants]
  Smokers | 7 | 5 | 12
  Non-Smokers | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinking Days
Description: Measured with time line follow back measures
Time Frame: 25 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Mecamylamine
Number analyzed (Participants) | 10 | 11
days | 17.6 (6.570) | 12.6 (6.570)
Statistical Analysis 1: Comparison: Placebo; Comparison is between baseline and during treatment; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — F=7.73

2. Primary Outcome: Depression - Measured Using the HAMD Total Score
Description: The Hamilton Depression Rating Scale (HAM-D) has proven useful for many years as a way of determining a patient's level of depression before, during, and after treatment. It should be administered by a clinician experienced in working with psychiatric patients.
  Although the HAM-D form lists 21 items, the scoring is based on the first 17. It generally takes 15-20 minutes to complete the interview and score the results. The Scale ranges from 0 (normal) to >23 (Very Severe Depression)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mecamylamine | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | 8.212 (1.592) | 8.10 (1.60)
Statistical Analysis 1: Comparison: Mecamylamine; Comparison of baseline and post-treatment; Test type: Superiority or Other; p = .0001, Mixed Models Analysis — F=36.32

3. Secondary Outcome: Mean Percentage of Number of Drinking Days by Smoking Status
Description: Two-way interaction between smoking and medication for percentage of drinking days captured by time line follow back surveys. Data are calculated as number of drinking days over the number of days in the study for smokers and nonsmokers receiving either mecamylamine or placebo.
Time Frame: 25 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Drinking Days
Arm/Group | Mecamylamine | Placebo
Number analyzed (Participants) | 11 | 10
Percentage of Drinking Days
  Smokers | 21.34 (21.96) | 4.57 (6.19)
  Non-Smokers | 14.76 (18.63) | 48.81 (35.22)
Statistical Analysis 1: Comparison: Mecamylamine vs Placebo; Test type: Superiority or Other; p = .025, Mixed Models Analysis

4. Secondary Outcome: Mean Percentage of Heavy Drinking Days by Smoking
Description: The two-way interaction between medication by smoking status to measure percentage of heavy drinking days measured by time line follow back survey. Data were calculated as number of heavy drinking days (heavy drinking days is defined as 5 drinks on a single occasion for men and 4 for women) over the number of days in the study for smokers and non smokers receiving either mecamylamine or placebo.
Time Frame: 25 weeks
Measure: Mean (Standard Deviation); unit: percentage of Heavy Drinking Days
Arm/Group | Mecamylamine | Placebo
Number analyzed (Participants) | 11 | 10
percentage of Heavy Drinking Days
  Smokers | 15.14 (19.48) | 1.68 (2.47)
  Non-Smokers | 3.57 (6.19) | 31.67 (29.03)
Statistical Analysis 1: Comparison: Mecamylamine vs Placebo; Test type: Superiority or Other; p = .019, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Placebo: Placebo capsules were prepared by the pharmacy and were identical in size and color to themedication capsules.
  Placebo: Placebo pill
Arm/Group | Mecamylamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 3/11 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mecamylamine (N=11) | Placebo (N=10)
Vomiting/Diarrhea (Gastrointestinal disorders) | 1 | 0
Relapse to Drinking (General disorders) | 1 | 1
Worsening of Depression (Psychiatric disorders) | 1 | 0
Calcified Granuloma (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes